CLINICAL TRIAL: NCT03034213
Title: Randomized, Controlled Trial Comparing Separation of Components Repair With Retrorectus Gentrix™ Surgical Matrix Versus Biological or Prosthetic Mesh for Open Ventral Hernia Repair
Brief Title: Gentrix™ Versus Biological or Prosthetic Mesh
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cease of Funding
Sponsor: University of South Florida (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA2017-002
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Ventral Incisional Hernia
Keywords: mesh
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Active Comparator): Gentrix(TM) Surgical Matrix
  Interventions: Device: Gentrix™ Surgical Matrix (Treatment)
- Control (Active Comparator): Standard of care mesh
  Interventions: Device: Permacol, Parietex, Progrip, Strattice Perforated, or Surgimend (Control)

INTERVENTIONS:
Device: Gentrix™ Surgical Matrix (Treatment) — Gentrix™ Surgical Matrix will be placed in the retrorectus space. The anterior midline fascia will be closed with long-acting absorbable suture either with a running or interrupted manner as per the surgeon's discretion.
  Arms: Treatment
Device: Permacol, Parietex, Progrip, Strattice Perforated, or Surgimend (Control) — A biological or prosthetic mesh (Permacol, Parietex, Progrip, Strattice Perforated, or Surgimend) will be placed in the retrorectus space. The anterior midline fascia will be closed with long-acting absorbable suture either with a running or interrupted manner as per the surgeon's discretion.
  Arms: Control

SUMMARY:
The hypothesis for this study is complex incisional hernia repair using the separation of components technique reinforced with retrorectus placement of Gentrix™ Surgical Matrix will lead to fewer incisional hernia recurrences and fewer wound complications compared to the same incisional hernia repair techniques reinforced with other prosthetic or biologically-derived mesh.

DETAILED DESCRIPTION:
Biological and prosthetic mesh products are extensively used in hernia repairs. However, they also have their limitations. Potential complications associated with prosthetic mesh for hernia repairs include: adverse reactions to the mesh, mesh erosion, stricture formation, adhesions resulting in bowel obstruction, enterocutaneous fistulas, injuries to nearby organs, nerves or blood vessels, infection, chronic pain and hernia recurrence. Potential complications associated with biological mesh include: adverse inflammatory response, laxity, eventration, and recurrent herniation. This study is a two-arm, randomized, controlled trial comparing separation of components repair with retrorectus Gentrix™ Surgical Matrix versus biological or prosthetic mesh for open ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years old.
* American Society of Anesthesiologists (ASA) physical status classification of I, II, III or IV.
* Able to provide informed consent in English or Spanish.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Body Mass Index (BMI) =< 45.
* Incisional hernia from a midline incision ≥ 4 cm in greatest diameter, or any recurrent incisional hernia.

Exclusion Criteria:

* Any other type of ventral hernia, such as umbilical, epigastric or Spigelian hernia.
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study, if applicable.
* Allergy or hypersensitivity to materials in porcine-based study products, biological or prosthetic meshes, or personal preference.
* Contraindications to general anesthesia.
* Patient undergoing any emergency surgery prior to treatment.
* Severe comorbid conditions likely to limit survival to less than 3 years in the opinion of the Investigator.
* Have abdominal loss of domain such that the operation would be impractical or would adversely affect respiratory or cardiovascular function to an unacceptable degree in the opinion of the Investigator.
* Inability to close the fascia primarily with abdominal wall mobilization or component separation; confirmed intra-operatively.
* History of malignancy within the past 5 years except for non-melanoma skin cancer.
* Known active malignancy present and/or had chemotherapy 12 weeks prior to screening or planned chemotherapy within 12 weeks of treatment with exception of basal cell carcinoma, squamous cell carcinoma, or prostate cancer in situ.
* Cirrhosis with or without ascites.
* Received high dose steroids (>/=100mg of prednisone) within the past 6 weeks of screening.
* Uncontrolled diabetes (i.e. known HbA1C value > 7% within the prior 6 weeks of the Screening Visit).
* History of drug addiction (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or the subject's ability to complete the required follow up.
* Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol.
* Suspected presence of enterocutaneous fistula.
* Planned use of external VAC dressing intra-operatively.
* Suspected bowel obstruction (partial or intermittent), strangulation, peritonitis, or perforation.
* Active necrotizing fasciitis or any other known active local or systemic infection.
* Subject report of participation in an investigational drug or device study that would impact the safety or scientific integrity of this study (in the opinion of the Investigator and with the approval of the Sponsor) within the past 6 weeks prior to treatment in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of incisional hernia recurrence | 2 years from study incisional hernia repair

SECONDARY OUTCOMES:
Time to incisional hernia recurrence | 2 years from study incisional hernia repair
Incidence of wound complications | 90 days from study incisional hernia repair
  Complications of interest: surgical site infections, seroma formation, and wound dehiscence or skin separation
Incidence of enterocutaneous fistula formation | 2 years from study incisional hernia repair
Mean Carolinas Comfort Scale score | 2 years from study incisional hernia repair
  Patient-centered outcome
Mean Visual Analog Scale score | 2 years from study incisional hernia repair
  Patient-centered outcome
Mean mesh deployment time | duration of surgery (incisional hernia repair)
  Defined as the time mesh preparation starts to time mesh placement ends
Mean procedure time | duration of surgery (incisional hernia repair)
  Defined as time of incision to time of closure
Mean total cost of hospitalization for primary admission | duration of hospitalization for incisional hernia repair
  Defined as from surgery to hospital discharge
Mean total cost of surgery for primary admission | duration of surgery (incisional hernia repair)
  Defined as from preoperative preparation to anesthesia discharge
Mean total cost of narcotic usage for primary admission | duration of hospitalization for incisional hernia repair
  Defined as narcotic use from surgery to hospital discharge
Mean total cost of readmissions | 2 years from study incisional hernia repair
  Defined as any hospital readmissions related to ventral hernia complications or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Vic Velanovich, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida
  - University of South Florida Morsani Center for Advanced Health Care, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FitzGerald JF, Kumar AS. Biologic versus Synthetic Mesh Reinforcement: What are the Pros and Cons? Clin Colon Rectal Surg. 2014 Dec;27(4):140-8. doi: 10.1055/s-0034-1394155. PMID 26106284
- [Background] Zhou XH, Melfi CA, Hui SL. Methods for comparison of cost data. Ann Intern Med. 1997 Oct 15;127(8 Pt 2):752-6. doi: 10.7326/0003-4819-127-8_part_2-199710151-00063. PMID 9382393
- [Result] Holihan JL, Alawadi Z, Martindale RG, Roth JS, Wray CJ, Ko TC, Kao LS, Liang MK. Adverse Events after Ventral Hernia Repair: The Vicious Cycle of Complications. J Am Coll Surg. 2015 Aug;221(2):478-85. doi: 10.1016/j.jamcollsurg.2015.04.026. Epub 2015 May 9. PMID 26206646
- [Result] Fekkes JF, Velanovich V. Amelioration of the effects of obesity on short-term postoperative complications of laparoscopic and open ventral hernia repair. Surg Laparosc Endosc Percutan Tech. 2015 Apr;25(2):151-7. doi: 10.1097/SLE.0000000000000100. PMID 25222715
- [Result] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861
- [Result] Fischer JP, Wink JD, Tuggle CT, Nelson JA, Kovach SJ. Wound risk assessment in ventral hernia repair: generation and internal validation of a risk stratification system using the ACS-NSQIP. Hernia. 2015 Feb;19(1):103-11. doi: 10.1007/s10029-014-1318-5. Epub 2014 Dec 4. PMID 25472771
- [Result] Heniford BT, Walters AL, Lincourt AE, Novitsky YW, Hope WW, Kercher KW. Comparison of generic versus specific quality-of-life scales for mesh hernia repairs. J Am Coll Surg. 2008 Apr;206(4):638-44. doi: 10.1016/j.jamcollsurg.2007.11.025. Epub 2008 Feb 1. PMID 18387468
- [Result] Nielsen K, Poelman MM, den Bakker FM, van der Ploeg T, Bonjer HJ, Schreurs WH. Comparison of the Dutch and English versions of the Carolinas Comfort Scale: a specific quality-of-life questionnaire for abdominal hernia repairs with mesh. Hernia. 2014 Aug;18(4):459-64. doi: 10.1007/s10029-013-1173-9. Epub 2013 Oct 29. PMID 24166693